CLINICAL TRIAL: NCT06335381
Title: Maternal OutcoMes (MOMs) Program: Testing Integrated Maternal Care Model Approaches to Reduce Disparities in Severe Maternal Morbidity
Brief Title: MOMs Chat and Care Study
Acronym: MOMs-CC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-0131; 1R01NR021134-01 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Severe Maternal Morbidity
Keywords: Maternal health; Severe maternal morbidity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups in parallel for the duration of the study.
Who Masked: Investigator
Masking Description: The Principal Investigator and Biostatistician will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOMs High Touch (MOMs-HT) (Experimental): Participants randomized to the MOMs-HT arm will receive close clinical and behavioral health monitoring via weekly chats (text or email) using chatbot technology and navigation to timely clinical, behavioral health, and/or social care services by the MOMs team throughout the prenatal and postpartum periods; 12 bi-weekly self-management support telehealth visits with a MOMs care management coordinator (CMC) or registered nurse (RN) during the prenatal period; home blood pressure monitor to measure their blood pressure regularly; Fitbit to track physical activity; and 5 bi-weekly telehealth visits with navigation to clinical, behavioral, and social services as needed by the MOMs team up to 6 weeks postpartum.
  Interventions: Other: Northwell Pregnancy & Peds Chats; Behavioral: Prenatal Telehealth Visits; Other: Postpartum Telehealth Visits; Other: Home Blood Pressure Monitor; Other: Fitbit
- MOMs Low Touch (MOMs-LT) (Active Comparator): Participants randomized to the MOMs-LT arm will receive close clinical and behavioral health monitoring via weekly chats (text or email) using chatbot technology and navigation to timely clinical, behavioral health, and/or social care services by the MOMs team throughout the prenatal and postpartum periods; 5 bi-weekly telehealth visits with navigation to clinical, behavioral, and social services as needed by the MOMs team up to 6 weeks postpartum; and a Fitbit to track physical activity.
  Interventions: Other: Northwell Pregnancy & Peds Chats; Other: Postpartum Telehealth Visits; Other: Fitbit

INTERVENTIONS:
Other: Northwell Pregnancy & Peds Chats — The Northwell Pregnancy & Peds Chats is a personalized care digital chatbot delivered via the Conversa platform. At Northwell, patients are enrolled automatically to receive the chats when they initiate prenatal care. Chats are accessible on a smartphone, tablet, and computer. During the prenatal and postpartum periods, participants receive a weekly chat via text message or email with a link to the platform. Each chat begins with asking if there are any updates the patient wants to share regarding their pregnancy. The chats provide timely, brief educational tools and resources. They are also designed to capture clinical, behavioral health, and social health concerns that triggers yellow flags (e.g., lack of transportation to obstetrics appointment) or red flags (e.g., elevated blood pressure) that go to a 24/7 nurse-led call center who follows up to connect the participant to clinical, behavioral health, or social services as needed.
Behavioral: Prenatal Telehealth Visits — The MOMs CMC/RN (interventionists) will deliver up to 12 bi-weekly self-management support telehealth visits during the prenatal period. The first telehealth visit will be 30-45 minutes in duration and follow-up visits will be 15-20 minutes. These telehealth visits will involve clinical and behavioral health check-ins; navigation to clinical, behavioral health, and social services as needed; screening for social needs during the initial telehealth visit; follow-up on referrals to resources to address social needs; and self-management support. MOMs CMCs/RNs will assess progress with engagement in self-management behaviors including asking about minutes and type of physical activity, self-monitoring (blood pressure, blood sugar, weight), and taking medications. The MOMs CMC/RN will provide brief maternal health education and support the participant in establishing behavior change goals and facilitating problem solving to address barriers to achieving goals each session.
  Arms: MOMs High Touch (MOMs-HT)
Other: Postpartum Telehealth Visits — The MOMs CMC/RN will conduct a telehealth visit (with navigation as needed) by phone 24 and 72 hours after labor and delivery. After the 72-hour call, telehealth visits with navigation will occur bi-weekly until 6 weeks postpartum. These telehealth visits will be 15-20 minutes in duration. Telehealth visits will include a brief clinical and behavioral health check-in, screening for social needs, navigation to clinical, behavioral health, and social services as needed, and follow-up on referrals to community resources and social services. During each visit, participants will be asked if they have experienced any signs or symptoms of concern (e.g., pain, discomfort, headaches, bleeding), screened for depression and anxiety, and be reminded about upcoming medical appointments. The CMC or RN will navigate the participant to the appropriate provider (e.g., OB, cardiologist, behavioral health) or services (e.g., emergency, social, community-based resources) as needed in a timely manner.
Other: Home Blood Pressure Monitor — Participants will receive an Omron 10 home blood pressure monitor to use throughout the study period. Along with the cuff, participants will receive written (postcard) and video instructions (https://youtu.be/p9UEDv6nvwU) on how to accurately measure their blood pressure. Participants with diagnosed chronic hypertension or preeclampsia during the prenatal period will be encouraged to measure their blood pressure twice a day; participants without these conditions will be encouraged to measure their blood pressure twice a week. During the postpartum period, participants will be encouraged to follow their provider recommendations in terms of how often they should measure their blood pressure. Participants will be allowed to keep the blood pressure monitor after the study has completed.
  Arms: MOMs High Touch (MOMs-HT)
Other: Fitbit — Participants will receive a Fitbit to use during the study period. Participants will be asked to wear the Fitbit on their wrist throughout the day to track all activity (e.g., walking, other physical activity, sedentary activity, and sleep). All data including minutes of activity and step counts will be stored on a secure web-based platform that aggregates data from the Fitbit device. Participants will be encouraged to sync their Fitbit device every 5 days with their phone to ensure data is up to date. Participants will be allowed to keep the Fitbit after the study has completed.

SUMMARY:
The purpose of this study is to test the effectiveness of an integrated care model approach at two different levels of intensity designed to facilitate timely, appropriate care to reduce risk for SMM. Black and Hispanic pregnant patients with an Obstetrics-Comorbidity Index Score ³ 2 and/or a history of pre-eclampsia will be identified via the electronic health record and 674 will be recruited and randomized early during pregnancy to one of two study arms: MOMs High-Touch (MOMs-HT) vs. MOMs Low-Touch (MOMs-LT). The two study arms will be compared on incidence of SMM at labor and delivery (Aim 1), incidence rate of SMM-related hospitalizations at 1-month and 1-year postpartum (Aim 1a), time to preeclampsia diagnosis and initiation of treatment (Aim 2), change in perceived social support domains (Aim 3), and physical activity trajectories (exploratory Aim 4). Mixed methods will also be used to examine facilitators and barriers to implementation (Aim 5). Findings from this study will help to determine how to feasibly implement an effective and sustainable integrated care approach to reduce risk for SMM.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of an integrated care model approach at two different levels of intensity designed to facilitate timely, appropriate care to reduce risk for SMM. Black and Hispanic pregnant patients with an Obstetrics-Comorbidity Index Score ³ 2 and/or a history of pre-eclampsia will be identified via the electronic health record and 674 will be recruited and randomized early during pregnancy to one of two study arms: MOMs High-Touch (MOMs-HT) vs. MOMs Low-Touch (MOMs-LT). MOMs-HT will consist of close clinical and behavioral health monitoring via chatbot technology and navigation to timely care and services by the MOMs team throughout the prenatal and postpartum periods; 12 bi-weekly self-management support calls with the MOMs team during the prenatal period; and 5 bi-weekly postpartum clinical check-in calls with navigation by the MOMs team up to 6 weeks postpartum. MOMs-LT will also include clinical and behavioral health monitoring via the chatbot along with navigation to services by the MOMs team as needed and 5 bi-weekly postpartum clinical check-in calls with navigation. Participants in both study arms will receive a Fitbit to track engagement in physical activity. SMM at labor and delivery (primary) and SMM-related hospitalizations at 1-month and 1-year postpartum (secondary) will be based on the CDC's 21 indicators with diagnoses extracted from the EHR. Diagnosis of preeclampsia and initiation of treatment (secondary) will also be captured using the EHR. Questionnaires will be administered to measure domains of social support (secondary). Physical activity behaviors (exploratory) will be assessed via survey and wearable activity monitor (i.e., Fitbit). Determinants of implementation will be captured via semi-structured qualitative interviews and discrete process measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older,
* Self-identify as Black/African American or Hispanic/Latina (includes Black + another race; Black or Afro Hispanic/Latina; or Hispanic/Latina),
* Pregnant, less than 17 weeks gestational age,
* OB-CMI risk score ≥ 2 and/or history or preeclampsia,
* English or Spanish as primary language, and
* Receive care at Northwell Health Physician Partners obstetrics practice site.

Exclusion Criteria:

• Birthing people who are not able to provide informed consent due to cognitive or psychiatric impairment.

If interested in participating in the study, please visit https://www.momschatandcare.com/

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 674 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe maternal morbidity (SMM) | Labor and delivery; 1-month postpartum; 1-year postpartum
  The Centers for Disease Control & Prevention define SMM as having ≥ 1 ICD-10 diagnosis codes that correspond to 21 SMM indicators. SMM indicator diagnoses that occur at labor and delivery, from delivery to 1-month postpartum during a hospital admission, or from delivery to 1-year postpartum during a hospital admission will be extracted from the electronic health record.

SECONDARY OUTCOMES:
Preeclampsia | During prenatal period (from study enrollment to labor and delivery), estimated 9 months.
  We will use the electronic health record to capture date preeclampsia diagnosis is documented at any time between study enrollment and labor and delivery (i.e., during the prenatal period) in both study arms. The following ICD-10 codes will be used to determine preeclampsia diagnosis: O14.1, O14.10, O14.12, O14.13, O14.14, or O14.15. Also, using the electronic health record and surveys, we will assess when treatment for preeclampsia (i.e., low-dose aspirin) has been initiated.
Informational Support | Baseline; 1-month postpartum; 1-year postpartum
  he PROMIS 10-item Informational Support measure will be administered to all participants to assess degree of support in terms of having someone to provide information or offer advice. The validated measure is on a 5-point Likert scale (ranging from 'never' to 'always') and is available in English and Spanish.
Emotional Support | Baseline; 1-month postpartum; 1-year postpartum
  The PROMIS 12-item Emotional Support measure will be administered to all participants to assess degree of feeling like they have someone who cares and expresses concern. The validated measure is on a 5-point Likert scale (ranging from 'never' to 'always') and is available in English and Spanish.
Tangible Support | Baseline; 1-month postpartum; 1-year postpartum
  This is a newly developed 8-item measure based on findings from qualitative interview with previous MOMs Program participants. The measure is designed to assess the degree to which patients feel supported in accessing clinical care and social services.

OTHER OUTCOMES:
Minutes of Physical Activity | Continuous (from enrollment to 1-year postpartum)
  Participants will be asked to wear the Fitbit during the entire study period. We will extract the total number of minutes of physical activity per week from the Fitbit for each participant.
Barriers to Exercise | Baseline; 1-month postpartum; 1-year postpartum
  The Barriers to Exercise Scale is a 14-item validated measure that will be administered to participants to assess barriers to engaging in exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Fitzpatrick, PhD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data related to the outcomes will be shared with scientists on the Open Science Framework (OSF) repository. This will include the 21 severe maternal morbidity indicators, preeclampsia diagnosis, and responses to the perceived social support domain measures. We will also include data relating to physical activity and data for variables which may moderate the primary analyses (e.g., sociodemographics, comorbidity). Data will be redacted to strip all individual identifiers, and effective strategies will be adopted to minimize risk of disclosing a participant's identity. Whenever possible, raw participant-level data will be shared along with documentation of how variables were cleaned, coded, or summarized. In cases where participant-level data could be used to identify individuals, summary data will be presented rather than raw data. Information about how summary data was generated will be provided in the data dictionary.
Supporting Information: Study Protocol
Time Frame: The intent is to make these data generally available, following the publication of the primary analyses of the study, and after the data have been appropriately checked, cleaned, and de-identified. Our expectation is that the data will be available within 9-12 months of the final year of funding. We will publicize the availability of the data after main results from the study have been published on both our Northwell website and presented at academic conferences.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to use the data only for research purposes, and not to identify any individual patient; 2) a commitment to secure the data using appropriate computer technology; and 3) a commitment to destroy or return the data after analyses are completed.

REFERENCES:
- [Derived] Fitzpatrick SL, Polo J, Ephraim P, Vrany E, Chiuzan C, Basile M, Friel CP, Moon KC, Silvia E, Bleau H, Nicholson W, Lewis D; MOMs Chat Care Research Group. MOMs Chat & Care Study: Rationale and design of a pragmatic randomized clinical trial to prevent severe maternal morbidity among Black birthing people. Contemp Clin Trials. 2025 May;152:107850. doi: 10.1016/j.cct.2025.107850. Epub 2025 Feb 21. PMID 39987957